CLINICAL TRIAL: NCT00166257
Title: Randomized Clinical Trial Comparing the Efficacy of Percutaneous Closure of Patent Foramen Ovale (PFO) With Medical Treatment in Patients With Cryptogenic Embolism
Brief Title: PC-Trial: Patent Foramen Ovale and Cryptogenic Embolism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Foundation for Cardiovascular Research, Zurich (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Meier, Bernhard, MD, Professor of Cardiology,, University of Berne, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICN98008
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2009-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Embolism, Paradoxical; Heart Septal Defects, Atrial
Keywords: Paradoxical embolism, Patent foramen ovale,
MeSH Terms: conditions — Embolism, Paradoxical; Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical antitrhombotic treatment (Active Comparator)
  Interventions: Drug: Medical antitrhombotic treatment
- Device Implant (Experimental): Percutaneous closure of patent foramen ovale
  Interventions: Device: Percutaneous closure of patent foramen ovale

INTERVENTIONS:
Device: Percutaneous closure of patent foramen ovale — Percutaneous implantation of an AMPLATZER® PFO Occluder
  Arms: Device Implant
Drug: Medical antitrhombotic treatment — Investigator's choice: Anticoagulation to INR 2.0 - 3.0 OR Aspirin 100-325 mg/d OR Clopidogrel 75-150 mg/d
  Arms: Medical antitrhombotic treatment

SUMMARY:
The purpose of this study is to compare two treatments strategies to prevent further attacks in patients who have suffered an stroke or occlusion of a major artery with no obvious reason other than a persistent small opening between the upper heart chambers

DETAILED DESCRIPTION:
In patients who have suffered a stroke or occlusion of a large artery in another body part of unknown origin a possible cause is a small opening between the upper heart chambers (patent foramen ovale, it is called). After birth this opening closes in 75% of the population, while it persists in 25% of people. It may allow a small blood clot to pass from the veins of the legs through the heart into the brain or other parts of the body. In order to reduce the risk for a further attack we have today more therapeutic options to choose from but it is unclear which strategy have the best outcome. This study is created to compare the effect of two treatment strategies:

1. Medical treatment The purpose of medical treatment is to dilute the blood to a degree, that no thrombus formation occurs. Since the opening in the heart persists, treatment is usually recommended lifelong. And patients treated with coumadin must undergo regular blood tests to ensure an adequate effect of the drug.
2. Catheter closure of patent foramen ovale An alternative method developed to close the small opening in the heart utilizes catheters which are introduced in a blood vessel in the groin and from there advanced to the heart. An umbrella device is then delivered through the catheter, positioned within the small defect and released. The umbrella is overgrown with own tissue within weeks to months and closes the small defect for ever.

ELIGIBILITY:
Inclusion Criteria:

* Age below 60 years
* Ischemic stroke or peripheral thromboembolism, radiologically verified
* Absence of an identifiable cause of embolism
* Echocardiographically verified patent foramen ovale
* Sufficient recovery from index event to allow independent daily activities

Exclusion Criteria:

* Any identifiable cause for thromboembolic event other than PFO
* Cardiac diseases: mural thrombus, dilated cardiomyopathy, prosthetic heart valve or mitral stenosis, endocarditis, atrial fibrillation
* Vascular system: significant atherosclerosis or dissection of the aorta, collagen vascular disease, arteritis, vasculitis
* Pre-existing neurologic disorders or intracranial disease, e.g., multiple sclerosis, arteriovenous malformations, previous hemorrhage
* Contraindications for antithrombotic or anticoagulant therapy
* Patients already on chronic anticoagulant therapy for another disease
* Previous surgical or percutaneous PFO-closure
* Drug or alcohol abuse
* Pregnancy
* Septicemia or severe infectious disease
* Severe CNS disease
* No informed consent
* Foreseen difficulties with study compliance, especially the long-term follow-up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 414 (Actual)
Dates: Start 2000-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Time to death (Fatal stroke, cardiovascular, non-CV), | continuosly
non-fatal cerebrovascular event, | continuosly
peripheral embolism | continuosly

SECONDARY OUTCOMES:
New arrhythmias, | continuosly
myocardial infarction | continuosly
rehospitalization related to PFO or its treatment | continuosly
device problems | continuosly
bleeding complications | continuosly

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Meier, MD, Study Chair — Dept. Cardiology, University Hospital Insel, Berne, Switzerland
Locations (6):
- Australia (3):
  - Monash Medical Centre, Melbourne
  - Sir Charles Gairdner Hospital, Nedlands
  - Alfred Hospital, Prahan
- Universitätsklinik für Innere Medizin II, Vienna, Austria
- A.Z. Sint-Jan AV, Bruges, Belgium
- University Hospital / Inselspital, Bern, Switzerland

REFERENCES:
- [Derived] Meier B, Kalesan B, Mattle HP, Khattab AA, Hildick-Smith D, Dudek D, Andersen G, Ibrahim R, Schuler G, Walton AS, Wahl A, Windecker S, Juni P; PC Trial Investigators. Percutaneous closure of patent foramen ovale in cryptogenic embolism. N Engl J Med. 2013 Mar 21;368(12):1083-91. doi: 10.1056/NEJMoa1211716. PMID 23514285
- [Derived] Khattab AA, Windecker S, Juni P, Hildick-Smith D, Dudek D, Andersen HR, Ibrahim R, Schuler G, Walton AS, Wahl A, Mattle HP, Meier B. Randomized clinical trial comparing percutaneous closure of patent foramen ovale (PFO) using the Amplatzer PFO Occluder with medical treatment in patients with cryptogenic embolism (PC-Trial): rationale and design. Trials. 2011 Feb 28;12:56. doi: 10.1186/1745-6215-12-56. PMID 21356042